CLINICAL TRIAL: NCT03483116
Title: A Phase II Randomized, Double Blind, Parallel Group Dose-ranging Study of Oral RV3-BB Rotavirus Vaccine Administered at a High, Mid and Low Titre as a 3 Dose Neonate Schedule or Administered at a High Titre as a 3 Dose Infant Schedule.
Brief Title: A Phase II Dose-ranging Study of Oral RV3-BB Rotavirus Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCRI-RV3-BB-004
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Rotavirus Infections
Keywords: Dose ranging; Neonatal vaccine; RV3-BB vaccine
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Intervention Model Description: This is a Phase II, randomised, double-blind, placebo-controlled, four-arm parallel group study of two different dosing schedules of oral RV3-BB
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- High dose RV3-BB neonatal schedule (Experimental): High dose neonatal RV3-BB vaccine schedule. RV3-BB Vaccine for Investigational product doses 1 (0-5 days), 2 (week 6) and 3 (week 10) and placebo for Investigational product dose 4 (week 14)
  Interventions: Biological: RV3-BB; Biological: Placebo
- Mid dose RV3-BB neonatal schedule (Experimental): Mid dose neonatal RV3-BB vaccine schedule. RV3-BB Vaccine for Investigational product doses 1 (0-5 days), 2 (week 6) and 3 (week 10) and placebo for Investigational product dose 4 (week 14)
  Interventions: Biological: RV3-BB; Biological: Placebo
- Low dose RV3-BB neonatal schedule (Experimental): Low dose neonatal RV3-BB vaccine schedule. RV3-BB Vaccine for Investigational product doses 1 (0-5 days), 2 (week 6) and 3 (week 10) and placebo for Investigational product dose 4 (week 14)
  Interventions: Biological: RV3-BB; Biological: Placebo
- High dose RV3-BB infant schedule (Experimental): High dose infant RV3-BB vaccine schedule. Placebo for Investigational product dose 1 (0-5 days) and RV3-BB Vaccine for Investigational product doses 2 (week 6) 3 (week 10) and dose 4 (week 14)
  Interventions: Biological: RV3-BB; Biological: Placebo

INTERVENTIONS:
Biological: RV3-BB — Oral administration
Biological: Placebo — Oral administration

SUMMARY:
The purpose of this study is to determine the serum IgA response of three dose levels of the oral RV3-BB vaccine when administered in a neonatal schedule or when administered as a high dose in an infant schedule.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the cumulative anti-rotavirus serum IgA response (defined as a ≥3 fold increase from baseline) 4 weeks after 3 doses of RV3-BB administered in a neonatal schedule at a High, Mid or low vaccine titre. In addition the cumulative anti-rotavirus serum IgA response (defined as a ≥3 fold increase from baseline) 4 weeks after 3 doses of RV3-BB administered in an infant schedule at a high dose of vaccine will be assessed along with cumulative vaccine take and components of vaccine take after 3 doses of RV3-BB administered in a neonatal or infant schedule.

The safety and tolerability of RV3-BB when administered as an infant or as a neonatal schedule will be described.

ELIGIBILITY:
Inclusion Criteria:

* Neonate is less than 6 days (≤144 hours) of age at the time of first dose.
* Neonate is in good health as determined by clinical judgment, including a medical history and physical exam, which confirms the absence of a current or past disease state considered significant by the investigator.
* Neonate birth weight 2500-4000g inclusive.
* Neonate's parents/guardians expect to be available for the duration of the study, and agree to adhere to all protocol requirements.
* Neonate's parents/guardians have provided written informed consent prior to study-related procedures being performed.

Exclusion Criteria:

* Any medical, psychiatric, or social condition of a parent/guardian that in the opinion of the investigator would prevent the neonate's parents/guardians from giving proper informed consent or from complying with the study protocol.
* Neonates with known or suspected major congenital malformations or genetically determined disease.
* Neonates with intussusception.
* Neonates with a known or suspected bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Neonates who have ever received any blood products, including immunoglobulin, or for whom receipt of any blood product during the course of the study is anticipated.
* Neonates in whom Essential Programme Immunisation (EPI) vaccines or components are contraindicated.
* Neonates who have received or who expect to receive during the study period, any rotavirus vaccine other than those which will be administered as part of this study.
* Neonates who have ever received, or who are anticipated to receive during the study period, any investigational agent other than those which will be administered as part of this study.
* Neonates with a previous anaphylactic reaction to any drug, vaccine or vaccine component.
* Neonates with a significant evolving neurological disorder.
* Neonates whose parents/guardians are site team employees with direct involvement with the investigators, or who are working on the study.
* Neonates who have been exposed to immunosuppressive courses of glucocorticosteroids, cytotoxic drugs or blood products through prenatal exposure and/or breast milk in the four weeks prior to randomization.
* Neonates with diarrhoea or vomiting in the 24 hours preceding randomisation.
* Neonates with any moderate or severe illness, and/or who have a temperature of ≥37.5˚C axillary/oral or ≥38˚C rectal/tympanic within the 48 hours preceding randomization.

Ages: 0 Days to 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 711 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Witte, MD MTropPaed, Principal Investigator — Malawi-Liverpool-Wellcome Trust Clinical Research Programme
Locations (1):
- Malawi-Liverpool-Wellcome Trust Clinical Research Programme, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified group data may be available for sharing on application to the Sponsor. This application must include the relevant proposal detailing the intended use of the data, the Ethics approval for this proposal and requires a signed data sharing agreement. Additional study documents including the study protocol, statistical analysis plan and informed consent are available on application to the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For 24 months from publication of the primary outcome.
Access Criteria: 1. Data access agreement
  2. Approval by local Ethics committee

REFERENCES:
- [Background] Witte D, Handley A, Jere KC, Bogandovic-Sakran N, Mpakiza A, Turner A, Pavlic D, Boniface K, Mandolo J, Ong DS, Bonnici R, Justice F, Bar-Zeev N, Iturriza-Gomara M, Ackland J, Donato CM, Cowley D, Barnes G, Cunliffe NA, Bines JE. Neonatal rotavirus vaccine (RV3-BB) immunogenicity and safety in a neonatal and infant administration schedule in Malawi: a randomised, double-blind, four-arm parallel group dose-ranging study. Lancet Infect Dis. 2022 May;22(5):668-678. doi: 10.1016/S1473-3099(21)00473-4. Epub 2022 Jan 20. PMID 35065683
- [Derived] Morgan B, Lyons EA, Handley A, Bogdanovic-Sakran N, Pavlic D, Witte D, Mandolo J, Turner A, Jere KC, Justice F, Ong DS, Bonnici R, Boniface K, Donato CM, Mpakiza A, Meyer A, Bar-Zeev N, Iturriza-Gomara M, Cunliffe NA, Danchin M, Bines JE. Rotavirus-Specific Maternal Serum Antibodies and Vaccine Responses to RV3-BB Rotavirus Vaccine Administered in a Neonatal or Infant Schedule in Malawi. Viruses. 2024 Sep 19;16(9):1488. doi: 10.3390/v16091488. PMID 39339964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A two-stage consent process was followed:
  * Pregnant women were invited to provide preliminary consent during the third trimester and prior to going into labour.
  * Post birth, the parents/guardians were invited to provide consent for their baby to participate in the study.
Period: Overall Study
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Started | 178 | 179 | 175 | 179
Completed | 150 | 156 | 149 | 148
Not Completed | 28 | 23 | 26 | 31
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 7
Not completed — Lost to Follow-up | 9 | 4 | 9 | 5
Not completed — Death | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 16 | 14 | 16
Not completed — Unknown other reason | 3 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule | Total
Number analyzed (Participants) | 178 | 179 | 175 | 179 | 711
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 178 | 179 | 175 | 179 | 711
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] — Age at first dose of investigational product Population: Full analysis Set (27 missing)
  Days
    number analyzed (Participants) | 170 | 173 | 169 | 172 | 684
    (all) | 1.4 (1.5) | 1.4 (1.42) | 1.4 (1.45) | 1.5 (1.39) | 1.5 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 84 | 88 | 96 | 369
  Male | 77 | 95 | 87 | 83 | 342
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 178 | 179 | 175 | 179 | 711
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 178 | 179 | 175 | 179 | 711

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Cumulative Anti Rotavirus Serum Immunoglobulin A (IgA) Response (≥3 Fold Increase From Baseline) in Neonatal Vaccine Schedule at High Mid and Low Dose of RV3-BB
Description: Cumulative anti rotavirus serum Immunoglobulin A (IgA) response is defined as a ≥3 fold increase from baseline at each serum collection time point to 4 weeks after 3 doses of RV3-BB
Time Frame: At serum collection at approximately 14 weeks of age
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule
Number analyzed (Participants) | 141 | 143 | 141
participants | 79 | 80 | 57
Statistical Analysis 1: Comparison: High Dose RV3-BB Neonatal Schedule vs Low Dose RV3-BB Neonatal Schedule; Test type: Non-Inferiority — Non-inferiority of the lower titre vaccine was demonstrated if the upper bound of the CI was below 20%; Response rate = 0.1553, 95% CI 2-sided [0.039 to 0.272]
Statistical Analysis 2: Comparison: High Dose RV3-BB Neonatal Schedule vs Mid Dose RV3-BB Neonatal Schedule; Test type: Non-Inferiority — Non-inferiority of the lower titre vaccine was demonstrated if the upper bound of the CI was below 20%; Response rate = 0.0010, 95% CI 2-sided [-0.115 to 0.117]
Statistical Analysis 3: Comparison: Mid Dose RV3-BB Neonatal Schedule vs Low Dose RV3-BB Neonatal Schedule; Non-inferiority of the lower titre vaccine was demonstrated if the upper bound of the CI was below 20%; Test type: Non-Inferiority — Non-inferiority of the lower titre vaccine was demonstrated if the upper bound of the CI was below 20%; Difference Response rate = 0.1543, 95% CI 2-sided [0.038 to 0.270]

2. Secondary Outcome: Number of Participants With a Cumulative Anti Rotavirus Serum IgA Response (≥3 Fold Increase From Baseline) After 3 Doses in an Infant RV3-BB Schedule
Description: Defined as a ≥3 fold increase from baseline to 4 weeks after 3 doses of RV3-BB at 18 weeks of age
Time Frame: At serum collection visit approximately 18 weeks of age
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 141 | 143 | 141 | 140
participants | 100 | 96 | 86 | 82

3. Secondary Outcome: Serum Anti Rotavirus IgA Titres in Participants Receiving RV3-BB in a Neonatal or Infant Schedule
Description: Expressed as geometric mean titres (GMTs) from baseline to post dose 3 of RV3-BB Minimum 10 Maximum 250,000 Higher score considered to be immunogenic.
Time Frame: At serum collection time points at approximately 14 and 18 weeks of age
Population: Per protocol
Measure: Geometric Mean (Standard Deviation); unit: geometric mean titres
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 141 | 143 | 141 | 140
geometric mean titres | 48.4 (22339.87) | 39.9 (21758.64) | 28.0 (7724.19) | 77.7 (25020.69)

4. Secondary Outcome: Number of Participants With a Cumulative "Vaccine Take" (Serum Anti Rotavirus IgA Response or Shedding of RV3-BB Vaccine Virus) and Components of Vaccine Take After 3 Doses of RV3-BB Administered in a Neonatal or Infant Schedule at a High Dose of RV3-BB.
Description: Vaccine take is defined as at least a threefold increase in serum anti-rotavirus immunoglobulin A (IgA) from baseline to post Investigational product dosing, or detectable RV3 shedding in stools (by ELISA or PCR) any day from day three to day five following administration of Investigational product. Cumulative vaccine take is defined as Vaccine take observed at the current assessment time point or following any previous dose
Time Frame: Sample collections at Week 0 through to approximately 14 and 18 weeks of age
Population: Per protocol analysis
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 141 | 140
participants
  Vaccine take | 118 | 120
  Serum IgA | 79 | 82
  Shedding RV3-BB vaccine virus | 85 | 90

5. Secondary Outcome: Number of Participants With Cumulative Vaccine Take and Components of Vaccine Take After 3 Doses of RV3-BB Administered in a Neonatal or Infant Schedule at a Mid or Low Dose of RV3-BB
Description: as for outcome 4
Time Frame: Sample collections at Week 0 through to approximately 14 and 18 weeks of age
Population: Per protocol analysis
Measure: Number; unit: participants
Arm/Group | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule
Number analyzed (Participants) | 143 | 141
participants
  Vaccine take | 114 | 94
  Serum IgA | 80 | 57
  RV3-BB Vaccine Shedding | 71 | 62

6. Secondary Outcome: Number of Participants With Cumulative Vaccine Take and Components of Vaccine Take After 2 Doses of RV3-BB Administered in a Neonatal or Infant Schedule at a High, Mid or Low Dose of RV3-BB
Description: as for outcome 4
Time Frame: Sample collections at Week 0 through to approximately 10 and 14 weeks of age
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 141 | 143 | 141 | 140
participants
  Vaccine take | 98 | 89 | 68 | 98
  Serum IgA | 56 | 55 | 31 | 58
  RV3-BB vaccine shedding | 69 | 52 | 46 | 70

7. Secondary Outcome: Number of Participants With Cumulative Vaccine Take and Components of Vaccine Take After 1 Dose of RV3-BB Administered in a Neonatal or Infant Schedule at a High, Mid or Low Dose of RV3-BB
Description: as for outcome 4
Time Frame: Sample collections at Week 0 through to approximately 6 and 10 weeks of age
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 141 | 143 | 141 | 140
participants
  Vaccine take | 51 | 45 | 23 | 64
  Serum IgA | 31 | 31 | 12 | 26
  RV3-BB vaccine shedding | 29 | 15 | 12 | 48

8. Secondary Outcome: Occurrence of Adverse Events (AE)
Description: Number of Participants with Adverse Events
Time Frame: First dose of investigational product to Study End at approximately 18 weeks of age
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 170 | 172 | 169 | 173
participants | 67 | 68 | 69 | 60

9. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs)
Description: Number of participants with Serious Adverse Events (SAEs)
Time Frame: First dose of investigational product to Study End at approximately 18 weeks of age
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 170 | 172 | 169 | 173
participants | 11 | 7 | 8 | 5

10. Secondary Outcome: Occurrence of Diarrhea. Severe
Description: Diarrhea will be described according to severity and detection of wild type rotavirus in diarrhea samples collected. Severity defined using a modified version of the Vesikari clinical score for gastroenteritis. Severed is modified Vesikari score of greater than or equal to 11.
  The Vesikari scale is a 20-point scale based on duration and peak frequency of diarrhea and vomiting, degree of temperature, severity of dehydration, and treatment provided to the patient (i.e., rehydration or hospitalization). This scale is divided into three ranges: mild <7, moderate 7-10, and severe ≥11
Time Frame: First dose of Investigational product to Study End at approximately 18 weeks of age
Population: Full analysis Set
Measure: Number; unit: participants
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
Number analyzed (Participants) | 178 | 179 | 175 | 179
participants | 1 | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: Adverse events were reported for the safety analysis set. The safety analysis set includes all randomised participants who received at least one dose of investigational product. Participants will be analysed according to the treatment received. Conditions identified as a congenital anomaly or birth defect, regardless of when the condition is identified, were not be recorded as SAEs unless the condition progressed/worsened or was fatal. These conditions were recorded as medical history.
Arm/Group | High Dose RV3-BB Neonatal Schedule | Mid Dose RV3-BB Neonatal Schedule | Low Dose RV3-BB Neonatal Schedule | High Dose RV3-BB Infant Schedule
All-Cause Mortality (participants affected / at risk) | 1/170 | 0/172 | 2/169 | 1/173
Serious Adverse Events (participants affected / at risk) | 11/170 | 7/172 | 8/169 | 5/173
Other Adverse Events (participants affected / at risk) | 67/170 | 68/172 | 69/169 | 59/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose RV3-BB Neonatal Schedule (N=170) | Mid Dose RV3-BB Neonatal Schedule (N=172) | Low Dose RV3-BB Neonatal Schedule (N=169) | High Dose RV3-BB Infant Schedule (N=173)
Bronchiolitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sepsis Neonatal (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Breast Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infantile Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose RV3-BB Neonatal Schedule (N=170) | Mid Dose RV3-BB Neonatal Schedule (N=172) | Low Dose RV3-BB Neonatal Schedule (N=169) | High Dose RV3-BB Infant Schedule (N=173)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 10 (12) | 9 (10) | 4 (5)
Bronchiolitis (Infections and infestations) | 8 (9) | 10 (10) | 6 (6) | 5 (6)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (5) | 8 (9) | 5 (5) | 7 (7)
Nasopharyngitis (Infections and infestations) | 11 (12) | 7 (8) | 5 (5) | 5 (5)
Opthalmia Neonatorum (Infections and infestations) | 4 (4) | 6 (6) | 3 (3) | 8 (8)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5) | 4 (4) | 1 (1)
Respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4) | 10 (10) | 4 (5)
Sepsis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3) | 1 (1)
Sepsis Neonatal (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
Upper Respiratory tract infection (Infections and infestations) | 15 (15) | 16 (16) | 16 (17) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 8 (8) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 6 (6) | 5 (5) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator must not Publish or present any aspect of the Study without the prior written approval of the Sponsor such approval will not to be unreasonably withheld

DOCUMENTS (2):
  • Study Protocol (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT03483116/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT03483116/SAP_001.pdf